CLINICAL TRIAL: NCT05979831
Title: A Phase 1b/2, Double-Blind, Placebo-Controlled, Randomized, Parallel-Arm Study to Explore Safety, Pharmacokinetics, and Early Clinical Signal of Efficacy of DS-2325a in Patients With Netherton Syndrome
Brief Title: A Study to Explore Safety, Pharmacokinetics, and Early Clinical Signal of Efficacy of DS-2325a in Patients With Netherton Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on a business decision by the Sponsor.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS2325-119; 2022-502853-32-00 (Other: EU CTR)
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Netherton Syndrome
Keywords: Netherton Syndrome; DS-2325a
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DS-2325a (Experimental): Participants will be randomized to receive a single initial ("loading") dose of DS-2325a (Week 1) followed by ("maintenance") doses for a total of 12 weeks (Main Phase).
  Participants will receive DS-2325 doses for a total of 24 weeks (Extension Phase).
  Interventions: Drug: DS-2325a
- Placebo (Placebo Comparator): Participants will be randomized to receive a single initial loading dose of placebo followed by maintenance doses of placebo for a total of 12 weeks (Main Phase).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DS-2325a — Main Phase and Extension Phase: Loading IV dose followed by maintenance SC doses
  Arms: DS-2325a
Other: Placebo — Main Phase: IV infusion followed by SC doses
  Arms: Placebo

SUMMARY:
Netherton Syndrome (NS) is a severe rare disease characterized by generalized scaling, erythema, and epidermal barrier defects. This study assessed the safety, pharmacokinetics (PK), and efficacy of DS-2325a in patients with NS.

DETAILED DESCRIPTION:
This study will explore the safety, pharmacokinetics (PK), and early clinical signal efficacy of DS-2325a in adult patients with NS. The primary objective of the study will be to explore the safety and tolerability of DS-2325a in patients with NS by administering DS-2325a for 12 consecutive weeks (Main Phase, which will be double-blind and during which some participants will receive placebo as a control) and to confirm by administering for an additional 24 weeks (Extension Phase, which will be open-label and during which all participants will receive DS-2325a). Secondary objectives of the study will include exploring the PK properties, efficacy, and immunogenicity of DS-2325a in patients with NS by administering DS-2325a for 12 consecutive weeks (Main Phase) and to confirm by administering for an additional 24 weeks (Extension Phase).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 65 years with clinical diagnosis of NS including at least 3 out of the 4 following clinical criteria:

  * Neonatal erythroderma
  * Bamboo hair and/or alopecia
  * Chronic atopy specified as food allergy and/or asthma and/or rhino-conjunctivitis and/or eczema for at least 2 years
  * Ichthyosis linearis circumflexa or scaling erythroderma or equivalent
* Immunohistochemistry documentation of absence of LEKTI in the skin or confirmed SPINK5 gene mutations
* NS involvement of ≥20% of Body Surface Area (BSA)
* Patients must give written informed consent to participation in the study prior to Screening
* Participants must be willing and able to understand and comply with study requirements
* Participants must be willing to have skin tape harvests collected from lesional and nonlesional skin areas

Exclusion Criteria:

* Any skin disease that may interfere with the diagnosis or evaluation of NS
* Any infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, or antifungals within 2 weeks before Screening visit
* Concomitant systemic disease not controlled by treatment. Stability for 3 months prior to Screening is required
* Kidney or liver disease with significant impairment of organ function (creatinine clearance <30 mL/min, calculated using the Cockcroft-Gault Equation, and Child-Pugh Class C; ALT and AST >2 × ULN range; total bilirubin >1 × ULN).
* Concomitant disease or condition that may interfere with, or treatment of which may interfere with, the conduct of the study or that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this study
* Any significant condition (eg, medical, psychiatric, or social) that according to Investigator's judgment would prevent compliance with study protocol and full study participation
* Known hypersensitivity to any ingredient of the study drug product
* Anticipation of the need for surgery or hospitalization during the study
* History of suicide attempt or suicidal ideation within 1 year prior to Screening
* History of substance abuse within 6 months prior to Screening or a positive urine drug test at Screening. Medical marijuana may be used per discretion of the Investigator
* History or positive test result for human immunodeficiency virus (HIV) at Screening
* Active hepatitis B virus (HBV) infection, determined by positive test result for hepatitis B surface antigen, at Screening
* Active hepatitis C virus (HCV) infection, determined as HCV ribonucleic acid (RNA) above the limit of detection in patients with positive HCV antibody titer, at Screening
* Use of topical drugs that may alter the course of NS (eg, topical corticosteroids and topical calcineurin inhibitors) within 2 weeks before Screening or anticipation of need to use these drugs during study drug
* Systemic treatment with corticosteroids, immunosuppressants, targeted therapeutics, biologics, and IV Ig within 8 weeks before Screening
* Participation in any other clinical study or expanded access program with an investigational drug or device within 4 weeks before Screening
* Suspected or confirmed COVID-19 within 4 weeks before or ongoing at Screening and planned vaccination against COVID-19 during study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events | Screening up to Week 45 (end of study)

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Trough Concentration (Ctrough) | Main Phase: Baseline and predose of Weeks 3, 5, 7, 9, and 11; Extension Phase: Predose of Weeks 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, 37, and 45
Mean Ichthyosis Area Severity Index (IASI) Scores | Screening; Observational: Predose of Weeks 1, 5, and 9; Main Phase: Baseline, predose of Weeks 3, 5, 7, 9, and 11; Extension Phase, predose of Weeks 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, and 37
  The IASI measures the severity of the erythema (IASI-Erythema) and scaling (IASI-Scaling) based on a 4-point Likert scale where 0 (none) and 4 (very severe). The total IASI is determined by adding IASI-Erythema and IASI-Scaling scores. Higher scores indicate worse clinical outcome.
Mean Investigator Global Assessment (IGA) Scores | Screening; Observational: Predose of Weeks 1, 5, and 9; Main Phase: Baseline, predose of Weeks 3, 5, 7, 9, and 11; Extension Phase, predose of Weeks 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, and 37
  The IGA measures, using a 5-point scale (0, clear; 1, almost clear; 2, mild; 3, moderate; 4, severe) erythema, scaling, inflammatory papules or plaques, oozing, and lichenification. Higher scores indicate worse clinical outcome.
Mean Itch Numerical Rating Scale (NRS) Scores | Screening; Observational: Predose of Weeks 1, 5, and 9; Main Phase: Baseline, predose of Weeks 3, 5, 7, 9, and 11; Extension Phase, predose of Weeks 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, and 37
  The Itch NRS is a self-rated single item scale designed for assessing worst pruritus in the past 7 days. The scale utilizes an 11-point NRS, scored from 0 (no itch) to 10 (worst imaginable itch. Higher scores indicate worse clinical outcome.
Skindex-29 Responses | Screening; Observational: Predose of Weeks 1, 5, and 9; Main Phase: Baseline, predose of Weeks 3, 5, 7, 9, and 11; Extension Phase, predose of Weeks 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, and 37
  The Skindex-29 is a self-reported measure of skin-related symptoms, functioning, and emotional well-being, designed for use across dermatologic conditions.
Dermatology Life Quality Index (DLQI) Questionnaire | Screening; Observational: Predose of Weeks 1, 5, and 9; Main Phase: Baseline, predose of Weeks 3, 5, 7, 9, and 11; Extension Phase, predose of Weeks 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, and 37
  The DLQI is a self-reported measure of patients' perception of the impact of skin diseases on different aspects of their quality-of-life over the last week.
Number of Participants With Anti-Drug Antibodies Against DS-2325a | Main Phase: Baseline and predose of Weeks 5 and 9; Extension Phase: Predose of Weeks 13, 17, 21, 25, 29, 33, 37, and 45

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Saint Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/